CLINICAL TRIAL: NCT06446583
Title: Study on the Impact of Preoperative Chewing Gum on Postoperative Nausea and Vomiting in Robotic Surgery
Brief Title: Preoperative Chewing Gum and Postoperative Nausea and Vomiting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Min Suk Chae (Other)
Responsible Party: Sponsor-Investigator, Min Suk Chae, Associate professor. CHAE, Min Suk, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KC24EISI0138
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative chewing gum group (Experimental): Upon arrival at the preoperative preparation room, patients begin chewing sugar-free gum provided by the preoperative nurse. They continue chewing until they enter the operating room (for at least 15 minutes). Before entering the operating room, it is confirmed that the gum has been discarded.
  Interventions: Other: Chewing sugar-free gum
- No preoperative chewing gum group (No Intervention): After arriving at the preoperative preparation room, patients wait without chewing gum until they enter the operating room.

INTERVENTIONS:
Other: Chewing sugar-free gum — Upon arrival at the preoperative preparation room, patients begin chewing sugar-free gum provided by the preoperative nurse. They continue chewing until they enter the operating room (for at least 15 minutes). Before entering the operating room, it is confirmed that the gum has been discarded.
  Arms: Preoperative chewing gum group

SUMMARY:
General anesthesia for surgery can often lead to postoperative nausea and vomiting (PONV). Additionally, decreased or paralyzed bowel movements are among the most common complications following abdominal surgery, causing pain, abdominal distension, nausea, and vomiting, which can delay patient recovery and extend hospital stays. Therefore, meticulous perioperative management is crucial.

In recent years, efforts have been made to reduce the burden of surgery, decrease postoperative complications, and promote rapid rehabilitation for a quicker return to daily life. These efforts also aim to reduce healthcare costs by shortening hospital stays and optimizing resources. Various interventions, such as early feeding, early removal of nasogastric tubes, and physical therapy, have been trialed in clinical settings to prevent prolonged bowel inactivity and paralysis. However, due to limited clinical efficacy, these methods are not routinely used.

Recently, many researchers have reported the benefits of chewing gum in enhancing bowel motility and reducing PONV. However, there is limited research on the impact of chewing gum on PONV in robotic surgeries, which are considered less invasive compared to open or laparoscopic surgeries. Furthermore, there is particularly scarce research on the effects of preoperative gum chewing.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 19 to under 70 years
2. Scheduled elective robotic surgery
3. American Society of Anesthesiologists (ASA) Physical Status Classification I or II

Exclusion Criteria:

1. Cases where robotic surgery was planned but suddenly converted to another type of surgery
2. Patients with a history of dental damage, dentures, loose or capped teeth, or other unstable dental conditions
3. Patients with a history of temporomandibular joint (TMJ) damage or surgery
4. Head and neck surgeries
5. Emergency surgeries
6. Refusal to participate in the study

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
nausea and vomiting | One hour after surgery, referring to the period spent in the post-anesthesia care unit
  Incidence of nausea and vomiting in the post-anesthesia care unit

IPD SHARING:
Plan to Share IPD: No